CLINICAL TRIAL: NCT05479058
Title: A Randomized, Double-blind, Controlled, Multi-center Study to Evaluate the Efficacy and Safety of Dose De-escalation of Orally Administered Filgotinib in Subjects With Ulcerative Colitis in Clinical Remission
Brief Title: A Study Evaluating the Effect of Filgotinib Dose De-escalation in Participants With Ulcerative Colitis (UC) in Remission
Acronym: CAPYBARA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: the planned number of participants needed to ensure adequate precision in the estimations and to draw meaningful conclusions was unlikely to be met, questioning the scientific value and ethical grounds for study continuation
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG0634-CL-341; 2022-000719-30 (EudraCT Number)
Record Dates: First submitted 2022-07-26; First posted 2022-07-29 (Actual); Results first posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — GLPG0634

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study was double-blinded to treatment assignment until the last subject has reached the primary analysis time point.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Filgotinib 200 mg (Experimental): Participants received filgotinib 200 mg and placebo to match filgotinib 100 mg once daily orally.
  Interventions: Drug: Filgotinib; Drug: Placebo
- Filgotinib 100 mg (Experimental): Participants received filgotinib 100 mg and placebo to match filgotinib 200 mg once daily orally.
  Interventions: Drug: Filgotinib; Drug: Placebo

INTERVENTIONS:
Drug: Filgotinib — Administered orally once daily
  Other Names: GS-6034; GLPG0634
Drug: Placebo — Administered orally once daily

SUMMARY:
Participants who were in clinical remission on 200 milligram (mg) filgotinib once daily for at least 2 consecutive quarterly visits in the ongoing SELECTION-LTE study (GS-US-418-3899, NCT02914535), were planned to be rolled over and randomized in this study. The primary objective of this study was to evaluate the efficacy of filgotinib in participants in stable clinical remission on 200 mg filgotinib once daily for whom the dose was decreased to 100 mg once daily compared to participants remaining on 200 mg once daily.

DETAILED DESCRIPTION:
Participants were planned to receive the blinded treatment until primary analysis time point. After unblinding at the study primary analysis time point, participants would have received unblinded treatment. The clinical trial was originally designed with the primary endpoint to be assessed at Week 48. Due to early termination of the study, none of the participants completed 48 weeks of treatment. All participants participated in blinded treatment period only and the study was unblinded globally after study completion.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants must have participated in the SELECTION-LTE study (GS-US-418-3899), who were on 200 mg filgotinib once daily and fulfilled the following conditions:

  * partial Mayo Clinical Score remission over a period of at least 2 consecutive quarterly visits in the SELECTION-LTE study (GS-US-418-3899) prior to screening of the present study;
  * free of corticosteroids for at least 12 weeks prior to and including baseline;
  * fecal calprotectin (FCP) ≤250 microgram per gram (μg/g) at last observation within 6 months prior to screening or FCP ≤250 μg/g during the screening of the present study.
  * sigmoidoscopy ES of 0 or 1 (local score) at screening.
* Willing to refrain from live attenuated vaccines during the study and for 12 weeks after the last dose of filgotinib in the study.
* Female participants of childbearing potential must have had a negative highly sensitive (serum beta human chorionic gonadotropin) pregnancy test during screening and must have agreed to continued monthly urine dipstick pregnancy testing during filgotinib treatment.
* Female participants of childbearing potential must have agreed to use highly effective contraception measures as defined in the protocol.

Key Exclusion Criteria:

* Any chronic medical condition (including but not limited to, cardiac or pulmonary disease, alcohol, or drug abuse) that, in the opinion of the investigator or sponsor, would make the participant unsuitable for the study or would prevent compliance with the study protocol.
* Participant had a known hypersensitivity to filgotinib ingredients or history of a significant allergic reaction to filgotinib ingredients as determined by the investigator.
* Female participant who was pregnant or breastfeeding, or intended to become pregnant or breastfeed, and/or plans to undergo egg donation or egg harvesting for the purpose of current or future fertilization, during the study and until the end of the study.
* Participant was unable or unwilling to comply with restrictions regarding prior and concomitant medication as described in the protocol.
* Participant had a positive QuantiFERON® tuberculosis (TB) test at screening or had 2 indeterminate QuantiFERON® TB test results that required Investigational product (IP) treatment interruption, or participant had sign and symptoms of TB reactivation at screening.
* History of malignancy during or in the last 5 years prior to participation in the UC parent studies, except for participants who had been successfully treated for nonmelanoma skin cancer or cervical carcinoma in situ.
* Participant met discontinuation criteria of the SELECTION-LTE study (GS-US-418-3899).

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2023-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galapagos Study Director, Study Director — Galapagos NV
Locations (50):
- United States (5):
  - University of Miami, Miami, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Gastro Center of Maryland - Columbia, Columbia, Maryland
  - Rapid City Medical Center, Rapid City, South Dakota
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
- Universitair Ziekenhuis Leuven Campus Gasthuisberg, Leuven, Belgium
- Czechia (2):
  - Hepato-Gastroenterology HK, Hradec Králové
  - GEP Clinic, Prague
- France (8):
  - CHU Amiens-Picardie, Amiens
  - Centre Hospitalier Universitaire Hôpital Nord Service D'Hépato-Gastro-Entérologie, Marseille
  - Centre Hospitalier Universitaire de Nantes Hôtel Dieu Service d'hépato-gastroentérologie, Nantes
  - Hôpital Haut-Lévêque Service d'Hépato-Gastro-Entérologie et Nutrition, Pessac
  - Centre Hospitalier Lyon Sud Service d'Hépato-Gastroentérologie, Pierre-Bénite
  - Hôpital Pontchaillou, Rennes
  - Hopital Nord - CHU de Saint-Etienne Service de Gastro-Entérologie, Saint-Etienne
  - Centre Hospitalier Universitaire de Nancy - Hôpital de Brabois Service d'Hépato-gastroentérologie, Vandœuvre-lès-Nancy
- Germany (5):
  - DRK KliniKlinik für Innere Medizin Schwerpunkt Gastroenterologieken Berlin Westend, Berlin
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - EUGASTRO GmbH, Leipzig
  - Klinikum Lüneburg, Lüneburg
  - Gastroenterologische Gemeinschaftspraxis Minden, Minden
- Hungary (2):
  - Dél-pesti Centrumkórház - Országos Hematológiai és Infektológiai Intézet, Budapest
  - Bugát Pál Kórház, Gyöngyös
- Italy (4):
  - IRCCS de Bellis Unità Operativa Complessa Gastroenterologia II, Castellana Grotte
  - Azienda Ospedaliero-Universitaria Mater Domini Unita Operativa Fisopatologia Digestiva, Catanzaro
  - Azienda Ospedaliero-Universitaria Pisana U.O. Gastroentrologia Stabilimento di Cisanello, Pisa
  - Istituto di Ricovero e Cura a Carattere Scientifico - Istituto Clinico Humanitas, Rozzano
- Poland (12):
  - Przychodnia Vitamed NFZ, Bydgoszcz
  - Gabinet Endoskopii Przewodu Pokarmowego, Krakow
  - Krakowskie Centrum Medyczne, Krakow
  - Centrum Opieki Zdrowotnej Orkan-Med, Ksawerów
  - Santa Familia - Centrum Badań Profilaktyki i Leczenia, Lodz
  - Gabinet Lekarski Dr. Hab. N. Med. Bartosz Korczowski, Rzeszów
  - Endoskopia Sopot, Sopot
  - Torunskiego Centrum Gastrologii I Endoskopii - Gastromed, Torun
  - H-T. Centrum Medyczne Spółka z Ograniczoną Odpowiedzialnością, Tychy
  - Niepubliczny Zakład Opieki Zdrowotnej VIVAMED Jadwiga Miecz, Warsaw
  - Bodyclinic, Warsaw
  - Centrum Medyczne Oporów, Wroclaw
- Mediclinic Panorama, Cape Town, South Africa
- South Korea (4):
  - Yeungnam University Medical Center, Daegu
  - Kyung Hee University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Yonsei University Health System Severance Hospital Gastroenterology, Seoul
- Hospital Universitario Virgen del Rocío, Seville, Spain
- National Taiwan University Hospital Center for Infection Control, Taipei, Taiwan
- United Kingdom (4):
  - Addenbrooke's Hospital, Cambridge
  - Norfolk and Norwich University Hospital, Norwich
  - Saint Helens and Knowsley Teaching Hospitals NHS Trust, Prescot
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were in clinical remission with filgotinib 200 milligrams (mg) once daily for at least 2 consecutive quarterly visits in the ongoing long-term extension (LTE) SELECTION-LTE study (GS-US-418-3899; NCT02914535) and who met the eligibility criteria, were rolled over and randomized to this study. Participants were enrolled at study sites in Poland, France, Germany, the United States, Belgium, Republic of Korea, Spain, and the United Kingdom.
Pre-assignment Details: The clinical trial was originally designed with the primary endpoint to be assessed at Week 48 after which participants would have received unblinded treatment. Due to early termination of the study, none of the participants completed 48 weeks of treatment. All participants participated in blinded treatment period only and the study was unblinded globally after study completion.
Period: Overall Study
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg
Started | 11 | 11
Completed | 0 | 0
Not Completed | 11 | 11
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Study terminated by sponsor | 10 | 10

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all randomized participants who were administered study drug at least once.
Groups:
- Total: Total of all reporting groups
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (8.5) | 58.3 (10.7) | 57.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 10 | 11 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 11 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Corticosteroid-free Clinical Remission Based on Modified Mayo Clinical Score (mMCS)
Description: The mMCS is a tool designed to measure disease activity for ulcerative colitis. The mMCS was calculated as the sum of the 3 subscores: stool frequency, rectal bleeding, and endoscopy. Each subscore was graded from 0 to 3 with higher scores indicating more severe disease activity. The total mMCS score ranged from 0 to 9 with higher scores indicating more severe disease activity.
  The mMCS remission was defined as a total score of score ≤2, with endoscopic subscore of ≤1, stool frequency subscore of ≤1, and a rectal bleeding subscore of 0.
  Corticosteroid-free mMCS remission was defined as being free of corticosteroids for at least 12 weeks.
Time Frame: Week 48
Population: As the study was terminated prior to any participant reaching the primary analysis time point at Week 48, the data for this endpoint was not collected and analyzed.
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Time to Patient-Reported Outcome Based on 2 Items (PRO2) Flare
Description: PRO2 flare was defined as a PRO2 score worsening of at least 2 points and an absolute PRO2 score of at least 3, with stool frequency subscore ≥2, and rectal bleeding subscore ≥1.
  PRO2 included items of stool frequency and rectal bleeding. The range of each item score was 0 to 3 with higher scores indicating more severe disease.
Time Frame: Baseline up to Week 48
Population: Participants in the Full Analysis Set (FAS) (all randomized participants who were administered study drug at least once) were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg
Number analyzed (Participants) | 11 | 11
days | NA [NA to NA] — Due to insufficient number of participants with PRO2 flare, the median and 95% CI data could not be calculated. | NA [NA to NA] — Due to insufficient number of participants with PRO2 flare, the median and 95% CI data could not be calculated.

3. Secondary Outcome: Time to ES-Confirmed UC Flare
Description: An ES-confirmed UC flare was defined as an increase in rectal bleeding subscore by at least 1 point and an increase in stool frequency subscore by at least 2 points and an increase in endoscopic subscore by at least 1 point. Each subscore graded from 0 to 3 with higher scores indicating more severe disease.
Time Frame: Baseline up to Week 48
Population: Participants in the FAS were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg
Number analyzed (Participants) | 11 | 11
days | NA [NA to NA] — Due to insufficient number of participants with ES-confirmed UC flare, the median and 95% CI data could not be calculated. | NA [NA to NA] — Due to insufficient number of participants with ES-confirmed UC flare, the median and 95% CI data could not be calculated.

4. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP)
Description: CRP is an acute-phase protein which provides an objective criterion of inflammatory activity.
Time Frame: Baseline, Week 4, Week 12, Week 24, Week 36, and Week 48
Population: Participants in the FAS with available data were analyzed. As the study was terminated prior to any participant reaching the Week 48 time point, the data for Week 48 time point was not collected and analyzed.
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg
Number analyzed (Participants) | 9 | 10
milligrams per liter (mg/L)
  Change at Week 4 | 0.166 (0.533) | 1.713 (4.423)
  Change at Week 12: number analyzed (Participants) | 6 | 7
  Change at Week 12 | 0.532 (1.128) | 10.406 (26.944)
  Change at Week 24: number analyzed (Participants) | 5 | 5
  Change at Week 24 | 0.156 (0.128) | 16.002 (34.093)
  Change at Week 36: number analyzed (Participants) | 3 | 3
  Change at Week 36 | 0.367 (0.192) | 1.443 (0.525)
  Change at Week 48: number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in Fecal Calprotectin (FCP)
Description: Fecal calprotectin, a very stable biomarker, was a 36 kilodalton calcium and zinc binding protein of S-100 protein family which was neutrophil derived. It represents 60% of cytosolic proteins in neutrophils and was a measurement of neutrophil migration to the gastrointestinal tract.
Time Frame: Baseline, Week 4, Week 12, Week 24, Week 36, and Week 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: milligrams per kilogram (mg/kg)
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg
Number analyzed (Participants) | 7 | 8
milligrams per kilogram (mg/kg)
  Change at Week 4 | -27.6 (37.2) | 142.5 (307.7)
  Change at Week 12: number analyzed (Participants) | 7 | 5
  Change at Week 12 | -16.7 (48.1) | 920.6 (1996.2)
  Change at Week 24: number analyzed (Participants) | 3 | 4
  Change at Week 24 | -52.0 (54.6) | 374.3 (674.8)
  Change at Week 36: number analyzed (Participants) | 2 | 3
  Change at Week 36 | -46.5 (65.8) | -8.0 (70.4)
  Change at Week 48: number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Score
Description: The IBDQ is disease-specific questionnaire used for an assessment of Health Related Quality of Life (HRQoL) in participants with the Inflammatory Bowel Disease (IBD). It comprised of 32 questions divided into four health subscales: bowel symptoms (10 questions); systemic symptoms, including sleep disorders and fatigue (5 questions); emotional function such as depression, aggression, and irritation (12 questions); and social function, meaning the ability to participate in social activities and to work (5 questions). The IBDQ total score was calculated as the sum of the responses (each ranging from 1 [severe problem] to 7 [normal health]) to all 32 questions. Total IBDQ score ranged from 32 to 224 with a higher score indicating a better HRQoL.
Time Frame: Baseline, Week 48
Population: As the study was terminated prior to any participant reaching the Week 48 time point, the data for this endpoint was not collected and analyzed.
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious Adverse Events (SAEs), and TEAEs Leading to Treatment Discontinuation
Description: An adverse event (AE) was any untoward medical occurrence, new or worsening of any preexisting condition, in a clinical study participant administered a medicinal product and which did not necessarily had to have a causal relationship with this treatment.
  A TEAE was defined as
  * An AE which had a start date equal to or after the date of the first administration of study drug in this study and no later than 30 days after last administration of study drug.
  * And was either a newly reported event, or a worsening of an existing event.
  Serious TEAE was defined as a TEAE that
  * Resulted in death and was life-threatening;
  * Required in-patient hospitalization or prolongation of existing hospitalization;
  * Resulted in persistent or significant disability/incapacity;
  * Was a congenital anomaly / birth defect;
  * Was medically significant.
Time Frame: Baseline up to Week 48
Population: Participants in the Safety analysis set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg
Number analyzed (Participants) | 11 | 11
Participants
  TEAEs | 6 | 6
  Serious TEAEs | 0 | 0
  TEAEs Leading to Treatment Discontinuation | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 48
Description: The Safety Analysis Set included all randomized participants who were administered study drug at least once.
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 6/11 | 6/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Filgotinib 200 mg (N=11) | Filgotinib 100 mg (N=11)
Gastroenteritis (Infections and infestations) | 1 | 1
Campylobacter infection (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Postmenopause (Social circumstances) | 0/8 | 1/6 — This is a sex-specific AE. Only female participants were at risk.

LIMITATIONS AND CAVEATS:
This study was terminated as the planned number of participants needed to ensure adequate precision in the estimations and to draw meaningful conclusions was unlikely to be met, questioning the scientific value and ethical grounds for study continuation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review and approve any results of the study or abstracts for professional meetings prepared by the investigator(s). Published data must not compromise the objectives of the study. Data from individual study centers in multicenter studies must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2023-03-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT05479058/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/58/NCT05479058/SAP_001.pdf